CLINICAL TRIAL: NCT02818595
Title: Development of Maternal Voice Recognition in Preterm Neonates
Acronym: PREMAVOIX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PI11-DR-WALLOIS
Record Dates: First submitted 2016-06-24; First posted 2016-06-30 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Infant, Premature
Keywords: voice recognition
MeSH Terms: conditions — Premature Birth | interventions — Electroencephalography

ARMS (2):
- Normal children (Experimental): Every child meet the age criteria and without ductus arteriosus persistence ultrasound or detectable neurological disorders after clinical, neurophysiological and radiological
  Interventions: Device: electroencephalogram (HR-EEG); Device: Near Infra Red Spectroscopy (NIRS)
- Abnormal children (Experimental): Every child meet the criteria of age and having a detectable neurological disease after clinical, neurophysiological and radiological as intraventricular hemorrhage .
  Interventions: Device: electroencephalogram (HR-EEG); Device: Near Infra Red Spectroscopy (NIRS)

INTERVENTIONS:
Device: electroencephalogram (HR-EEG)
Device: Near Infra Red Spectroscopy (NIRS)

SUMMARY:
Many cognitive functions in humans are based on asymmetrical brain networks. For example, in most adults, the language is essentially processed by the left hemisphere, while other auditory functions, such as voice recognition, tend to be processed by the right hemisphere. Many studies, especially those conducted by Ghislaine Dehaene's team, have demonstrated the presence of anatomical and functional asymmetries by the first months of life. What are the causes of these asymmetries? How do they develop? Are they necessary for functioning or effective learning?

This study, conducted in collaboration with the Compiègne applied mathematics team (Abdelatif El Badia) and the INSERM team (Ghislaine Dehaene), is designed to determine the stage of development at which hemispheric dominance for voice recognition is first observed and to identify the brain structure involved in preterm neonates whose sound environment is usually very different from that of the foetus. The impact of this environment on the infant's brain development and early learning will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* The distribution of children in the different groups of infants included in the study will be validated at the time of the acquisitions.
* Normal group of children: A child meets the age criteria and without ductus arteriosus persistence ultrasound or detectable neurological disorders after clinical, neurophysiological and radiological (ETF, Scanner, MRI).
* Group of children meet the age criteria and with cerebral neurological pathology detectable after clinical, neurophysiological and radiological (ETF, Scanner, MRI).

Exclusion Criteria:

About history:

* All children with severe congenital malformation

Regarding the study period;

* Any refusal of a parent
* Children with severe impairment of the general condition and vital functions
* Children with dermatitis of the face or scalp
* Children treated with ventilation High Frequency (HFO)
* Presence of intravenous access on the scalp (preventing the realization of the ETF, EEG and NIRS

Ages: 0 Days to 6 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2013-03; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
The difference in amplitude | 10 weeks
  The difference in amplitude of the electrical hemodynamic responses to stimuli depending on the conditions, which corresponds to the evoked potential mismatch Response
The difference in latency | 10 weeks
  The difference in latency of the electrical hemodynamic responses to stimuli depending on the conditions, which corresponds to the evoked potential mismatch Response

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice WALLOIS, MD, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

REFERENCES:
- [Result] Beauchemin M, Gonzalez-Frankenberger B, Tremblay J, Vannasing P, Martinez-Montes E, Belin P, Beland R, Francoeur D, Carceller AM, Wallois F, Lassonde M. Mother and stranger: an electrophysiological study of voice processing in newborns. Cereb Cortex. 2011 Aug;21(8):1705-11. doi: 10.1093/cercor/bhq242. Epub 2010 Dec 13. PMID 21149849